CLINICAL TRIAL: NCT00005801
Title: A Phase II Study of Allografting to Establish Mixed or Full Donor Chimerism as Consolidative Immunotherapy for Older Patients With AML in Complete Remission Using Low Dose TBI, PBSC Infusion and Post-Transplant Immunosuppression With Cyclosporine and Mycophenolate Mofetil
Brief Title: Total-Body Irradiation Plus Stem Cell Transplantation And White Blood Cell Infusion in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 00-0119; UCHSC-00119; FHCRC-1406.00; NCI-G00-1778
Record Dates: First submitted 2000-06-02; First posted 2004-04-12 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2001-09

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); adult acute monocytic leukemia (M5b)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by radiation therapy used to kill tumor cells. Infusions of donor white blood cells may decrease the body's rejection of the transplanted peripheral stem cells.

PURPOSE: Phase II trial to study the effectiveness of combining radiation therapy, peripheral stem cell transplantation, and donor white blood cell infusions in treating older patients who have acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether mixed or full donor chimerism can be safely established in older patients with acute myeloid leukemia (AML) treated with nonmyeloablative conditioning comprised of low dose total body irradiation, followed by allogeneic peripheral blood stem cell transplantation, followed by unrelated donor lymphocyte infusion (DLI). II. Determine whether mixed chimerism can be safely converted to full donor chimerism in patients treated with DLI. III. Determine the potential efficacy of this regimen in AML patients who are in first remission.

OUTLINE: Conditioning: Patients undergo low dose total body irradiation followed by infusion of allogeneic peripheral blood stem cells (PBSC) on day 0. Donor lymphocyte infusions: Nonmobilized donor lymphocytes are harvested from the same HLA identical related donor on day 95 after PBSC transplantation. Eligible patients with mixed chimerism and no graft versus host disease (GVHD) receive the first donor lymphocyte infusion (DLI) on the same day that donor lymphocytes are collected. Patients who continue to have mixed chimerism and no GVHD receive the second DLI at a higher dose level on day 65 after the first DLI. Patients are followed weekly until day 90, and then monthly thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myeloid leukemia (AML) (de novo or secondary, FAB M1, M2 and M4-7) Must be within 6 months of diagnosis Achieved a chemotherapy induced first complete remission (CR) Received 1 or more courses of consolidation chemotherapy OR AML in second or greater CR Patients with a documented first or subsequent CR may proceed to transplantation if: No morphologic diagnosis of AML or myelodysplastic syndrome Absolute neutrophil count greater than 1,000/mm3 and platelet count greater than 50,000/mm3 after any consolidation chemotherapy Availability of an HLA identical related peripheral blood stem cell donor No syngeneic donor No active CNS leukemia

PATIENT CHARACTERISTICS: Age: Over 55 to under 75 Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) ALT and AST less than 4 times ULN Renal: Creatinine clearance at least 50 mL/min Cardiovascular: Cardiac ejection fraction at least 40% No poorly controlled hypertension Pulmonary: No severe defects in pulmonary function testing No requirement for supplementary continuous oxygen

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter McSweeney, MD, Study Chair — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Denver, Colorado
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241